CLINICAL TRIAL: NCT03803514
Title: Effect of Recombinant Erythropoietin in Plasma Levels of FGF23 in End-Stage Renal Disease Patients
Brief Title: Effect of rEPO in FGF23 in ESRD Patients
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Luis Toro, Co-researcher, University of Chile
Other Study IDs: ID-11102-23
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Anemia; Chronic Kidney Diseases
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated group (rEPO): Patients with ESRD in HD, and medical indication of recombinant EPO for management of anemia (Hb < 10 g/dL). Ambulatory hemodialysis 3 times per week.
  Recombinant beta-epoetin (Recormon) will be used, according to current recommendations.
  Clinical and laboratory data will be obtained before and during the study. The primary outcome (changes of plasma intact FGF23) will be measured during the follow-up, up to 12 weeks.
  Interventions: Drug: Recombinant EPO
- Control group: Patients with ESRD and HD, without medical indication of recombinant EPO (Hb > 10 g/dL). Ambulatory hemodialysis 3 times per week.
  Follow-up for 3 months, similar than rEPO group. Clinical and laboratory data will be obtained before and during the study, similar periods than rEPO group.
  The primary outcome (changes of plasma FGF23) will be measured every 2 week during the evaluation period.

INTERVENTIONS:
Drug: Recombinant EPO — Beta-epoetin (Recormon, Roche). Dosage was performed according to current recommendations.
  Other Names: rEPO
  Groups: Treated group (rEPO)

SUMMARY:
Objective: To evaluate the effects of recombinant Erythropoietin (rEPO) in plasma levels of Fibroblast Growth Factor 23 (FGF23) in End-Stage Renal Disease (ESRD) patients in hemodialysis.

Method: Prospective cohort of ESRD patients in HD, where patients with or without rEPO therapy were compared. Measurements of plasma FGF23 were performed at baseline and during the complete study. Demographic, clinical and laboratory data will be obtained.

Follow-up period: 12 weeks.

DETAILED DESCRIPTION:
Experimental data has shown that recombinant erythropoietin (rEPO) increases plasma levels of Fibroblast Growth Factor 23 (FGF23) in murines, both health and with acute or chronic renal disease. Also, observational studies indicate an association between EPO and FGF23 levels in patients. Until now, it has not been demonstrated whether the use of rEPO does increase plasma FGF23 in End-Stage Renal Disease (ESRD) patients in hemodialysis (a population with a high use of this therapy for the management of chronic anemia).

Our objective was to evaluate whether the administration of rEPO increases plasma FGF23 levels in ESRD patients in hemodialysis.

We performed a prospective cohort with ESRD patients without rEPO therapy. We performed 2 groups: patients with requirements of rEPO therapy due to anemia (Hb < 10 g/dL) and patients without rEPO therapy (Hb > 10 g/dL).

We measured plasma FGF23 (intact and C-terminal) at baseline and during 12 weeks.

Demographic, clinical and laboratory data was obtained. Patients treated with rEPO received beta-epoetin (Recormon, Roche), according to current recommendations.

Patients were follow-up during 3 months to evaluate the effects of rEPO. Our primary outcome was changes in plasma intact FGF23 at 12 weeks, between both groups.

ELIGIBILITY:
Inclusion Criteria:

* End-Stage Renal Disease
* Requirements of Hemodialysis
* At least 6 months since initiation of hemodialysis

Exclusion Criteria:

* Pregnancy
* Treatment with rhEPO or analogs during the previous 6 months or earlier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pacients in chronic hemodialysis, will be measured with FGF23 levels
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Changes in plasma intact FGF23 levels | 12 weeks
  Measurements of plasma intact FGF23 levels

SECONDARY OUTCOMES:
Changes in plasma C-terminal FGF23 levels | 12 weeks
  Measurements of plasma C-terminal FGF23 levels
Changes in hematocrit and hemoglobin | 12 weeks
  Measurements of hematocrit and hemoglobin in blood samples
Changes in parathormone levels | 12 weeks
  Measurements of parathormone levels in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Luis Michea, MD PhD, Study Chair — University of Chile
Locations (1):
- Hospital Clinico Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided